CLINICAL TRIAL: NCT03669718
Title: A Randomized, Double-blind, Placebo-Controlled, Phase 2 Study of Cemiplimab Versus the Combination of Cemiplimab With ISA101b in the Treatment of Subjects With HPV16-Positive Oropharyngeal Cancer (OPC)
Brief Title: A Randomized Phase 2 Study of Cemiplimab ± ISA101b in HPV16-Positive OPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ISA Pharmaceuticals (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISA101b-HN-01-17
Record Dates: First submitted 2018-08-11; First posted 2018-09-13 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Squamous Cell Carcinoma of the Oropharynx; HPV16 Positive
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — cemiplimab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active ISA101b and cemiplimab. (Experimental): ISA101b 3 times plus cemiplimab every 3 weeks for up to 24 months
  Interventions: Biological: ISA101b; Drug: Cemiplimab
- Placebo and cemiplimab (Placebo Comparator): Placebo 3 times plus cemiplimab every 3 weeks for up to 24 months
  Interventions: Drug: Cemiplimab; Other: Placebo

INTERVENTIONS:
Biological: ISA101b — Every 3 weeks for a total of 3 times
  Arms: Active ISA101b and cemiplimab.
Drug: Cemiplimab — Every 3 weeks for up to 24 months
Other: Placebo — Every 3 weeks for a total of 3 times
  Arms: Placebo and cemiplimab

SUMMARY:
This will be a blinded, placebo-controlled, randomized, phase 2 study in which subjects will be randomly assigned 1:1 to cemiplimab plus placebo or cemiplimab plus ISA101b.

DETAILED DESCRIPTION:
This study will assess the ability of ISA101b to improve Overall Response Rate in subjects with HPV16 positive OPC, when combined with cemiplimab, an investigational anti-PD-1 antibody being developed by Regeneron Pharmaceuticals. ISA101b is a therapeutic cancer vaccine that induces specific immune responses to the oncogenic E6 and E7 antigens from HPV16. Trials in HPV16 driven malignancies indicate it has activity in HPV16 driven malignancies including oropharyngeal and cervical cancers. Cemiplimab, also known as REGN2810, is in late stage trials and appears to have similar activity to approved anti PD-1 antibodies in a number of malignancies .

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ≥ 18 years of age.
* Sign and date an Institutional Review Board/Independent Ethics Committee (IRB)/(IEC)-approved written informed consent form (ICF) in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal subject care.
* Be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study.
* Diagnosed with histologically confirmed recurrent or metastatic HPV16 positive OPC, whose tumors express PD-L1 (Combined Positive Score [CPS] ≥1) and who are candidates for first line therapy with an PD-1 blocking antibody, AND subjects with recurrent or metastatic HPV16 positive OPC with disease progression on or after platinum containing chemotherapy.
* HPV-16 genotyping will be determined by the specified central reference laboratory.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST 1.1 criteria.
* Prior curative radiation therapy must have been completed at least 4 weeks prior to study drug administration. Prior focal palliative radiotherapy must have been completed at least 2 weeks before study drug administration.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of study drug.

Exclusion criteria:

* Subjects with previously untreated metastatic or unresectable, recurrent HPV16 positive OPC whose tumors do not express PD-L1 (CPS<1) and who are therefore not candidates for monotherapy with an anti-PD-1 antibody.
* Subjects with known brain metastases or leptomeningeal metastases.
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
* History of other malignancy ≤ 3 years prior to entry into this trial with the exception of basal cell or squamous cell skin carcinoma which were treated with local resection only, or carcinoma in situ of the cervix, prostate or breast, or low grade non-muscle invasive superficial bladder cancer (TaLG)/carcinoma in situ of the bladder.
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Subjects with a condition requiring immunosuppressive doses of systemic medication such as steroids or absorbed topical steroids (doses ≥ 10 mg/day prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses < 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Prior treatment with an anti-PD-1 antibody (e.g., nivolumab, pembrolizumab, cemiplimab), as well as an antibody targeting anti-PL-L1 anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co stimulation or immune checkpoint pathways.
* Prior treatment with more than one chemotherapy regimen for the management of metastatic OPC.
* Prior treatment with therapeutic anti-HPV vaccines including ISA101 or ISA101b. Subjects may have received a preventive HPV vaccine.
* All toxicities attributed to systemic prior anti-cancer therapy other than alopecia and fatigue must have resolved to Grade 1 (NCI CTCAE) or baseline before administration of study drug. Subjects with toxicities attributed to systemic prior anticancer therapy that are not expected to resolve and result in long lasting sequelae, such as neuropathy after platinum based therapy, are permitted to enroll.
* History of allergy to ISA101/ISA101b study drug components, e.g., ISA101/101b, Montanide, or Macrogolglycerol Ricinoleate, also known as cremophore.
* History of allergy to cemiplimab and its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2018-11-30 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 25months
  Measured using RECIST 1.1
Number of participants with treatment-related adverse events as assessed by NCI CTCAE v5.0 "Number of participants with treatment-related adverse events as assessed by NCI CTCAE v5.0". | 25 months

SECONDARY OUTCOMES:
Duration of response (DOR) by independent review in subjects randomized to receive ISA101b plus cemiplimab compared to placebo plus cemiplimab. | 25months

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie S. Glisson, MD, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (44):
- United States (10):
  - City of Hope, Duarte, California
  - Moores Cancer Center at the UC San Diego Health, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - ICAHN School of Medicine at Mount Sinai, New York, New York
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - M. D. Anderson Cancer Center, Houston, Texas
- University Hospital Antwerp, Antwerp, Belgium
- Brazil (2):
  - DFSATR/Oncologia D'Or, Brasília
  - Instituto do Cancer do Estado de Sao Paulo, São Paulo
- Czechia (2):
  - University Hospital Olomouc, Olomouc
  - Nemocnice na Bulovce, Prague
- France (5):
  - Centre Léon Bérard, Lyon
  - CHU La Timone, Marseille
  - Antoine Lacassagne Center, Nice
  - Gustave Roussy, Paris
  - Hopitaux Universitaires Pitié Salpêtrière Charles Foix, Paris
- Universitaetsklinikum Ulm, Ulm, Germany
- Hungary (3):
  - Szabolcs Szatmar Bereg Megyei Korhazak Es Egyetemi Oktatokorhaz, Nyíregyháza
  - University of Pecs Department of Oncotherapy, Pécs
  - Hetenyi Geza Korhaz-Rendelointezet, Szolnok
- Italy (5):
  - ASST Spedali Civili Brescia, Department of Medical Oncology, Brescia
  - Azienda Ospedaliera San Paolo Polo Universitario, Milan
  - Istituto Nazionale dei Tumori, Milan
  - National Cancer Institute - IRCCS "Fondazione G. Pascale", Naples
  - National Cancer Institute Regina Elena, IRCCS, Rome
- Consultorio de Oncología Médica, Oaxaca City, Mexico
- Netherlands (3):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Radboud University Medical Center, Nijmegen
  - University Medical Center Utrecht, Utrecht
- Poland (2):
  - Maria Sklodowska-Curie National Institute of Oncology, Gliwice
  - Swietokrzyskie Oncology Center Kielce, Kielce
- Spain (4):
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital Duran i Reynals - Institut Catala dOncologia ICO, Barcelona
  - Vall d'Hebron, Barcelona
  - Hospital Universitario Marqués de Valdecilla Santander, Santander
- United Kingdom (5):
  - Aberdeen Royal Infirmary, Aberdeen
  - The Royal Marsden NHS Foundation, Chelsea
  - Guy's Hospital, London
  - The Royal Marsden NHS Foundation Trust, Sutton
  - Beacon Centre Musgrove Park Hospital, Taunton

REFERENCES:
- [Derived] Even C, Harrington KJ, Massarelli E, Laban S, Fayette J, Oliva M, Klein Hesselink M, Visscher S, Fury MG, Wiekmeijer AS, Licitra L, Melichar B, Devriese LA, Brana I, Jankowska P, Posner M, Glisson B, Kong A, Hooftman L, Melief CJM MD,, Ferrarotto R. Randomized clinical efficacy and safety study of peltopepimut-S plus cemiplimab compared to cemiplimab alone in patients with recurrent/metastatic HPV16-positive head and neck cancer. J Immunother Cancer. 2025 Sep 8;13(9):e012555. doi: 10.1136/jitc-2025-012555. PMID 40921630